CLINICAL TRIAL: NCT00314561
Title: The Effect of Pioglitazone and Rosiglitazone on Atherosclerotic and Inflammatory Markers in Patients With Metabolic Syndrome: A Prospective, Randomized, Open-label, Crossover Trial
Brief Title: The Effect of Pioglitazone and Rosiglitazone on Atherosclerotic and Inflammatory Markers in Patients With Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KoreaUAnanmH
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2008-09

CONDITIONS: Metabolic Syndrome
Keywords: Rosiglitazone; Pioglitazone; FMD; PWV; atherosclerosis
MeSH Terms: conditions — Metabolic Syndrome; Atherosclerosis | interventions — Pioglitazone; Rosiglitazone

INTERVENTIONS:
Drug: Pioglitazone, Rosiglitazone

SUMMARY:
Pioglitazone and rosiglitazone are used in the treatment of diabetic patients. Thiazolidinediones increase insulin sensitivity and show favorable effect blood glucose levels and lipid profiles. The effect of these two different thiazolidinediones on atherosclerotic and inflammatory markers has not been compared in prospective manner. The purpose of this prospective, randomized, open-label, crossover trial is to compare the effect of pioglitazone and rosiglitazone on atherosclerotic and inflammatory markers in patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 3 metabolic syndrome criteria of Asian-Pacific ATP III guideline: fasting blood glucose ≥ 110 mg/dl, systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 85 mmHg, triglyceride ≥ 150 mg/dl, HDL-cholesterol < 40 mg/dl for men and < 50 mg/dl for women.
* Age: 18 years and above

Exclusion Criteria:

* Hypertensive patients with the use of ACE inhibitor or ARB
* Hyperlipidemic patients with the use of statin or fenofibrate
* Patients with any contraindications to the treatment of thiazolidinediones
* Pregnant or lactating patients
* Chronic alcohol or drug abuse
* Hepatic dysfunction
* Renal dysfunction
* Heart failure (EF < 50%)
* Expected life expectancy of < 1 year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-05; Study Completion 2006-12

PRIMARY OUTCOMES:
The effect on flow-mediated dilation (FMD) and pulse wave velocity (PWV)

SECONDARY OUTCOMES:
The effect of atherosclerotic and inflammatory markers such as adiponectin, IL-6, TNF-α, hsCRP.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Sup Choi, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, Seoul, South Korea